CLINICAL TRIAL: NCT00266032
Title: A Multicenter, Open, Randomized, Parallel Group Comparison to Assess the Safety and Efficacy of the Oral Contraceptive SH T00186D (0.02 mg Ethinylestradiol as Betadex Clathrate and 3 mg Drospirenone) in Two Variations of an Extended Regimen vs. a Standard Regimen (24 + 4 Days) in 1122 Healthy Female Volunteers for One Year, Followed by a One Year Safety Extension
Brief Title: Study on Safety and Efficacy of an Oral Contraceptive in Long Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91450; 2005-002125-32 (EudraCT Number); 308683 (Other: Company Internal)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Contraception
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flexible (extended) treatment of EE20/DRSP (YAZ, BAY86-5300) (Experimental): 3 cycles of treatment, each cycle comprising 120 days intended treatment with one tablet daily of 20µg ethinyl estradiol as betadex clathrate (EE20) plus 3 mg drospirenone (DRSP) followed by a 4 day tablet-free interval. If 3 consecutive days of bleeding and/or spotting occurred during the 120 day treatment period, a 4 day tablet free interval was advised. The minimum period between 2 tablet free intervals was 24 days. After each 4 day tablet free interval, a new 120 day intended treatment period was to be restarted, resulting in a minimum of 3 and maximum of 13 withdrawal bleeding episodes during one year of treatment.
  Interventions: Drug: Flexible (extended) treatment of EE20/DRSP (YAZ, BAY86-5300)
- Fixed extended treatment of EE20/DRSP (YAZ, BAY86-5300) (Experimental): 3 cycles of treatment, each cycle comprising 120 days uninterrupted treatment with one tablet daily of 20µg ethinyl estradiol as betadex clathrate plus 3 mg drospirenone followed by a 4 day tablet free interval, 3 withdrawal bleeding episodes during one year of treatment were expected.
  Interventions: Drug: Fixed extended treatment of EE20/DRSP (YAZ, BAY86-5300)
- Standard 24+4 treatment of EE20/DRSP (YAZ, BAY86-5300) (Active Comparator): 13 cycles of treatment, each cycle comprising an intake of one tablet daily with 24 days of active tablets (20µg ethinyl estradiol as betadex clathrate plus 3 mg drospirenone) followed by 4 days of placebo tablets, 13 withdrawal bleeding episodes during one year of treatment were expected.
  Interventions: Drug: Standard 24+4 treatment of EE20/DRSP (YAZ, BAY86-5300)

INTERVENTIONS:
Drug: Flexible (extended) treatment of EE20/DRSP (YAZ, BAY86-5300) — 3 cycles of treatment, each cycle comprising 120 days intended treatment with one tablet daily of 20µg ethinyl estradiol as betadex clathrate (EE20) plus 3 mg drospirenone (DRSP) followed by a 4 day tablet-free interval. If 3 consecutive days of bleeding and/or spotting occurred during the 120 day treatment period, a 4 day tablet free interval was advised. The minimum period between 2 tablet free intervals was 24 days. After each 4 day tablet free interval, a new 120 day intended treatment period was to be restarted, resulting in a minimum of 3 and maximum of 13 withdrawal bleeding episodes during one year of treatment.
  Arms: Flexible (extended) treatment of EE20/DRSP (YAZ, BAY86-5300)
Drug: Fixed extended treatment of EE20/DRSP (YAZ, BAY86-5300) — 3 cycles of treatment, each cycle comprising 120 days uninterrupted treatment with one tablet daily of 20µg ethinyl estradiol as betadex clathrate plus 3 mg drospirenone followed by a 4 day tablet free interval, 3 withdrawal bleeding episodes during one year of treatment were expected.
  Arms: Fixed extended treatment of EE20/DRSP (YAZ, BAY86-5300)
Drug: Standard 24+4 treatment of EE20/DRSP (YAZ, BAY86-5300) — 13 cycles of treatment, each cycle comprising an intake of one tablet daily with 24 days of active tablets (20µg ethinyl estradiol as betadex clathrate plus 3 mg drospirenone) followed by 4 days of placebo tablets, 13 withdrawal bleeding episodes during one year of treatment were expected.
  Arms: Standard 24+4 treatment of EE20/DRSP (YAZ, BAY86-5300)

SUMMARY:
The purpose of the study is to determine safety and efficacy of long-cycle regimens of an oral contraceptive.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG (BSP AG), Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

The previously posted secondary Outcome Measure "Parameters of safety and tolerability" has been removed from result posting as it is covered by the Adverse Event section.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women who desire contraception
* smokers ≤ 30 Years old

Exclusion Criteria:

* Contraindication against use of hormonal contraceptives

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1166 (Actual)
Dates: Start 2005-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- Canada (6):
  - Drummondville, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Shawinigan, Quebec
  - Ste-Foy, Quebec
- Germany (20):
  - Ettlingen, Baden-Wurttemberg
  - Karlsruhe, Baden-Wurttemberg
  - Ansbach, Bavaria
  - Krumbach, Bavaria
  - Nuremberg, Bavaria
  - Hamburg, Hamburg
  - Dietzenbach, Hesse
  - Frankfurt am Main, Hesse
  - Mühlheim am Main, Hesse
  - Bovenden, Lower Saxony
  - Hanover, Lower Saxony
  - Osnabrück, Lower Saxony
  - Wurzen, Saxony
  - Bernburg, Saxony-Anhalt
  - Jessen, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Gera, Thuringia
  - Jena, Thuringia
  - Kahla, Thuringia
- Groningen, Netherlands

REFERENCES:
- [Result] Klipping C, Duijkers I, Fortier MP, Marr J, Trummer D, Elliesen J. Long-term tolerability of ethinylestradiol 20 mug/drospirenone 3 mg in a flexible extended regimen: results from a randomised, controlled, multicentre study. J Fam Plann Reprod Health Care. 2012 Apr;38(2):84-93. doi: 10.1136/jfprhc-2011-100214. PMID 22454004
- [Result] Klipping C, Duijkers I, Fortier MP, Marr J, Trummer D, Elliesen J. Contraceptive efficacy and tolerability of ethinylestradiol 20 mug/drospirenone 3 mg in a flexible extended regimen: an open-label, multicentre, randomised, controlled study. J Fam Plann Reprod Health Care. 2012 Apr;38(2):73-83. doi: 10.1136/jfprhc-2011-100213. PMID 22454003
- [Result] Reif S, Snelder N, Blode H. Characterisation of the pharmacokinetics of ethinylestradiol and drospirenone in extended-cycle regimens: population pharmacokinetic analysis from a randomised Phase III study. J Fam Plann Reprod Health Care. 2013 Apr;39(2):e1-13. doi: 10.1136/jfprhc-2012-100397. PMID 23493606
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization scheme in the subgroups was 1:1:1 for the 2 centers performing biopsies and measurements of Bone Mineral Density and metabolic parameters (82 subjects per treatment group). The remaining subjects were randomized according to the ratio 4:1:1.
Pre-assignment Details: 146 subjects failed screening, 96 of these 146 (65.8%) because inclusion or exclusion criteria were not met, 21 (14.4%) due to withdrawal of consent, 17 (11.6%) because of "other" reasons, 11 (7.5%) due to protocol deviations, 1 (0.7%) was lost to follow-up. 32 randomized subjects never took medication.
Period: Treatment
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Started | 691 (all randomized subjects, baseline data for full analysis set (FAS) only) | 236 (all randomized subjects, baseline data for full analysis set (FAS) only) | 239 (all randomized subjects, baseline data for full analysis set (FAS) only)
Patients Treated | 684 | 221 | 229
Patients Treated and in FAS | 642 (FAS) | 209 (FAS) | 216 (FAS)
Completed | 580 (not all entered period 2 (open-label safety extension)) | 172 (not all entered period 2 (open-label safety extension)) | 192 (not all entered period 2 (open-label safety extension))
Not Completed | 111 | 64 | 47
Not completed — Adverse Event | 42 | 26 | 10
Not completed — Lost to Follow-up | 19 | 4 | 2
Not completed — Pregnancy | 3 | 2 | 2
Not completed — Protocol Violation | 6 | 14 | 13
Not completed — Withdrawal by Subject | 28 | 13 | 12
Not completed — patient moved/wish for pregnancy/no need | 13 | 5 | 8
Period: Open-label Safety Extension
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Started | 489 (treatment for subjects of all 3 treatment groups in 2nd period, except for 28 in subgroups) | 129 (7 subjects continued their treatment in second period (safety extension)) | 165 (21 subjects continued their treatment in second period (safety extension))
Completed | 448 | 115 | 140
Not Completed | 41 | 14 | 25
Not completed — Adverse Event | 5 | 0 | 4
Not completed — Lost to Follow-up | 2 | 5 | 4
Not completed — Pregnancy | 4 | 1 | 2
Not completed — Protocol Violation | 1 | 3 | 2
Not completed — Withdrawal by Subject | 19 | 3 | 12
Not completed — patient moved/wish for pregnancy/no need | 10 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300) | Total
Number analyzed (Participants) | 642 | 209 | 216 | 1067
Age, Continuous [Mean (Full Range); unit: years] — Number of Participants analyzed for baseline was Full Analysis Set (FAS=safety set)
  years | 24.8 [18 to 35] | 24.8 [18 to 35] | 24.3 [18 to 35] | 24.7 [18 to 35]
Sex: Female, Male [Count of Participants; unit: Participants] — Number of Participants analyzed for baseline was Full Analysis Set (FAS=safety set)
  Participants
    Female | 642 | 209 | 216 | 1067
    Male | 0 | 0 | 0 | 0
Body-Mass-Index (BMI) [Mean (Full Range); unit: kg/m²] — Body mass index was calculated with body weight and height measured at screening (BMI = body weight in kg²/ body height in m³) and had to be 18 Years to 35 Years old (smokers ≤ 30 Years old) at inclusion.
  Number of Participants analyzed for baseline was Full Analysis Set (FAS=safety set).
  kg/m² | 22.541 [17.95 to 30.50] | 22.541 [18.00 to 29.70] | 22.566 [17.90 to 29.80] | 22.546 [17.90 to 30.50]

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Bleeding Including Spotting
Description: The number of bleeding days per volunteer was calculated by summing up all days with bleeding intensity spotting or worse. The primary evaluation was the comparison of the flexible extended vs the standard regimen for this primary target variable, which was done for data within the first year of treatment only. As no further comparison or testing was done, no multiplicity issue arose.
Time Frame: up to 1 year
Population: Full Analysis Set (FAS) (reflecting Intention To Treat (ITT) population), all treated subjects with data available, no imputation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 640 | 209 | 215
days | 41 (29) | 61 (51) | 66 (27)
Statistical Analysis 1: Comparison: Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) vs Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300); Primary variable was tested for the hypothesis, whether the means are equal against the alternative (means are different) at a level of significance of alpha = 0.05 (t-test). For power calculation, a normal distribution, a absolute difference of 10 days, a Standard Deviation of 28 days and a drop-out rate of 40% was assumed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -25, 95% CI [-29 to -20], Standard Deviation 29 — Mean of Yaz flexible regimen minus mean of Yaz standard was tested

2. Primary Outcome: Number of Unintended Pregnancies in Yaz Flexible Arm
Description: Pregnancies with conception date within 4 days after end of study medication were regarded as during treatment.
Time Frame: up to 2 years
Population: Full Analysis Set (reflecting ITT population), all treated subjects, no imputation, including switchers to flexible treatment in second year
Measure: Number; unit: pregnancies
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 879
pregnancies | 8

3. Primary Outcome: Pearl Index
Description: The Pearl Index (PI) is defined as the number of pregnancies per 100 woman years. The 2-year PI was obtained by dividing the number of pregnancies that occurred during the two years of treatment by the time (in 100 women years) that the women were under risk of getting pregnant. 95% confidence interval according to European Medicine Agency Note for guidance on clinical investigation of steroid contraceptives in women.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Pregnancies per 100 woman years
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 879
Pregnancies per 100 woman years | 0.64 [0.28 to 1.26]

4. Primary Outcome: Number of Unintended Pregnancies Due to Method Failure
Description: Not included in this analysis are pregnancies due to subject failure eg. non-compliance with tablet intake rules.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Number; unit: Pregnancies
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 875
Pregnancies | 7

5. Primary Outcome: Adjusted Pearl Index
Description: The adjusted Pearl Index was based on pregnancies due to method failures and compliant treatment cycles, i.e. cycle length between 24 and 124 day, pill break not longer than 7 days, and number of pills taken not smaller than 90% of the number of days in that cycle minus 7 days.
Time Frame: Up to 2 years
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Pregnancies per 100 woman years
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 875
Pregnancies per 100 woman years | 0.60 [0.24 to 1.24]

6. Secondary Outcome: Number of Days With Bleeding Excluding Spotting
Description: The number of bleeding days per volunteer was calculated by summing up all days with bleeding intensity light, normal, or heavy.
Time Frame: up to 1 year
Population: FAS
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 640 | 209 | 215
Days | 21 (15) | 24 (24) | 43 (20)

7. Secondary Outcome: Number of Bleeding Days During One Year of Treatment in Subjects With at Least 248 Days of Exposure Normalized to 372 Days
Description: For early dropouts and pregnant subjects with an exposure period of less than 1 year but at least 248 days, the number of bleeding/spotting days was normalized to correspond to a 1-year exposure period.
Time Frame: up to 1 year
Population: FAS (reflecting ITT population), all treated subjects, no imputation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 563 | 168 | 189
Days | 44 (29) | 66 (55) | 71 (24)

8. Secondary Outcome: Number of Bleeding / Spotting Days by 90-day Reference Period
Description: The mean number of bleeding / spotting days, spotting-only and bleeding days was analyzed using reference periods of 90 days as recommended by the WHO.
Time Frame: up to 1 year
Population: FAS (reflecting ITT), all treated subjects, no imputation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 605 | 182 | 203
Days
  Reference period 1 | 7.2 (5.5) | 9.0 (8.6) | 14.6 (6.1)
  Reference period 2 | 5.3 (5.6) | 6.3 (6.5) | 10.2 (4.8)
  Reference period 3 | 4.6 (4.3) | 5.1 (5.8) | 9.8 (4.8)
  Reference period 4 | 3.9 (4.5) | 2.6 (5.6) | 9.5 (4.9)

9. Secondary Outcome: Number of Bleeding / Spotting Episodes in 90 Day Reference Period
Description: The mean number of bleeding / spotting episodes was analyzed using reference periods of 90 days as recommended by the WHO.
Time Frame: Up to one year
Population: FAS (reflecting ITT), all treated subjects, no imputation
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 605 | 182 | 203
Episodes
  Reference period 1 | 1.7 (1.7) | 2.0 (1.9) | 3.4 (1.2)
  Reference period 2 | 1.9 (1.5) | 2.1 (1.4) | 3.4 (1.1)
  Reference period 3 | 1.7 (1.5) | 2.1 (1.8) | 3.2 (1.0)
  Reference period 4 | 1.5 (1.5) | 1.3 (1.5) | 3.2 (1.0)

10. Secondary Outcome: Days With Scheduled Versus Unscheduled Bleeding
Description: Days with scheduled and unscheduled bleeding were evaluated for extended regimens only. Unscheduled is any bleeding/spotting that occurred while taking active hormones regardless of the duration of intake, unless they occurred after tablet-free interval during days 1-4 of subsequent treatment cycle, or unless they occurred during days 1-7 of first treatment cycle. Scheduled is any bleeding/spotting that occurred during tablet-free interval, regardless of duration of tablet intake, or during next 4 days of subsequent treatment cycle.
Time Frame: Up to one year
Population: FAS (reflecting ITT), all treated subjects, no imputation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 640 | 209
Days
  Scheduled bleeding | 23.3 (14.3) | 14.0 (5.9)
  Unscheduled bleeding | 17.1 (17.4) | 46.6 (48.4)

11. Post Hoc Outcome: Number of Unintended Pregnancies Including Pregnancies Occuring Within 14 Days After End of Study Medication.
Description: Pregnancies with conception date during treatment and within 14 days after end of study medication were included.
Time Frame: Up to one year
Population: FAS
Measure: Number; unit: Pregnancies
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 639
Pregnancies | 2

12. Post Hoc Outcome: Pearl Index (FDA Criteria)
Description: Following an FDA request another PI evaluation was done for the first year of treatment only and taking into consideration also pregnancies with a conception date within 14 days after end of the study medication. Restricting the analysis to the required first year of treatment, it results in this PI estimation.
Time Frame: Up to one year
Population: FAS
Measure: Mean (95% Confidence Interval); unit: Pregnancies per 100 woman years
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 639
Pregnancies per 100 woman years | 0.34 [0.04 to 1.23]

ADVERSE EVENTS:
Arm/Group | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300)
Serious Adverse Events (participants affected / at risk) | 19/642 | 7/209 | 3/216
Other Adverse Events (participants affected / at risk) | 310/642 | 116/209 | 121/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) (N=642) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) (N=209) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300) (N=216)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gynaecological chlamydia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic peritoneal adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flexible (Extended) Treatment of EE20/DRSP (YAZ, BAY86-5300) (N=642) | Fixed Extended Treatment of EE20/DRSP (YAZ, BAY86-5300) (N=209) | Standard 24+4 Treatment of EE20/DRSP (YAZ, BAY86-5300) (N=216)
Abdominal pain lower (Gastrointestinal disorders) | 14 (14) | 12 (12) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 60 (82) | 24 (31) | 22 (28)
Nausea (Gastrointestinal disorders) | 27 (34) | 11 (12) | 12 (18)
Vomiting (Gastrointestinal disorders) | 36 (52) | 12 (15) | 9 (12)
Fatigue (General disorders) | 20 (25) | 7 (8) | 13 (15)
Influenza like illness (General disorders) | 13 (19) | 14 (21) | 18 (22)
Cystitis (Infections and infestations) | 33 (46) | 23 (32) | 14 (20)
Gastroenteritis (Infections and infestations) | 34 (38) | 15 (17) | 13 (14)
Influenza (Infections and infestations) | 23 (29) | 10 (13) | 14 (16)
Nasopharyngitis (Infections and infestations) | 129 (213) | 43 (62) | 53 (83)
Sinusitis (Infections and infestations) | 17 (22) | 13 (17) | 11 (12)
Vulvovaginal candidiasis (Infections and infestations) | 25 (36) | 12 (14) | 12 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 12 (13) | 13 (14)
Headache (Nervous system disorders) | 88 (168) | 41 (62) | 48 (76)
Dysmenorrhoea (Reproductive system and breast disorders) | 31 (41) | 11 (12) | 15 (22)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 9 (12) | 11 (17)

LIMITATIONS AND CAVEATS:
Data for center no. 1148 was included in "all randomized" set of subjects, but not in FAS, as during medical monitoring of laboratory data a suspicion of potential misconduct was found. An audit was made, but the suspicion could not be resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bayer Schering Pharma (BSP AG) coordinates publishing of study results. Principal investigators (PIs) provide BSP AG with a draft at least 90 days prior to date of planned submission or presentation. BSP AG shall have 60 days to recommend any changes. BSP AG can prevent or delay publication by informing PIs within 60 days of BSP AG´s receipt of the document about to be published. PIs shall not publish press releases/other public statements about study/study drug without BSP AG´s written consent.